CLINICAL TRIAL: NCT05274919
Title: Vascular Signature Mapping of Brain Tumor Genotypes
Acronym: VASIM
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Matthias van Osch, Prof. Dr. Ir. Matthias van Osch, Leiden University Medical Center
Other Study IDs: VSMBTG
Record Dates: First submitted 2022-02-08; First posted 2022-03-11 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Glioma
Keywords: MR imaging
MeSH Terms: conditions — Glioma | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients scheduled for brain MRI with contrast injection: Inclusion at Erasmus MC and LUMC: The first cohort consists of 60 patients scheduled for brain MRI as part of their standard clinical diagnostic procedure and in whom contrast agent administration is part of their standard radiological assessment. These patients do not necessarily have a brain tumor as the purpose here is to develop and evaluate the vascular signature mapping sequence in general. Usually, such testing would be done in healthy volunteers, but contrast agent is required for the vascular signature mapping sequence. To avoid unnecessary contrast agent administration, the sequence will be tested in this patient cohort instead. In this study part, the outcome is the optimized protocol itself, with which the investigators could obtain additional information about the vascular structure throughout the brain. Therefore this group of subjects is expected to be sufficiently homogeneous for the research aim of this part of the study.
  Interventions: Device: X-ray (optional); Other: Question list
- Patients diagnosed with suspected glioma scheduled for brain MRI: Inclusion at Erasmus MC and LUMC: The second cohort consists of 20 glioma patients in whom the vascular signature mapping sequence is tested specifically for glioma and for a direct comparison between 3T and 7T, where the 3T scan is an extension of the diagnostic care and the additional 7T scan is optional. This number of patients is sufficient to provide information on differences in the ability to measure tumor vascularity between 3T and 7T, while minimizing the extra patient burden.
  Interventions: Device: Philips Achieva 7T MRI; Device: X-ray (optional); Combination Product: Additional contrast injection; Other: Question list
- Patients with (suspected) glioma: Inclusion at Erasmus MC and LUMC: The third cohort consists of 100 adult patients referred for biopsy or surgery of suspected glioma. The diagnosis of glioma is based on a multitude of factors, such as initial presentation (headaches, vomiting, potential changes in character). Based on the initial presentation a patient may be suspected of having a glioma, which is often confirmed using imaging. Although a true conclusion requires analysis of tissue, in an overwhelming majority of the cases (99%), analysis of the imaging is sufficient to confirm the presence of glioma. Thus, the investigators can be relatively certain about the inclusion of glioma patients based on the initial presentation and imaging alone.
  Since there is a close collaboration with the Neurology departments of both the LUMC and Haaglanden Medical Center (HMC) in The Hague, the investigators broaden their inclusion capacity also to this hospital.
  Interventions: Device: Philips Achieva 7T MRI; Device: X-ray (optional); Combination Product: Additional contrast injection; Other: Question list

INTERVENTIONS:
Device: Philips Achieva 7T MRI — Regular follow-up MRI on 3T scanner and optional additional scan at 7T MRI.
  Other Names: Philips Ingenia (Elition) 3T MRI; GE Healthcare (MR750/Signa Premier) 3T MRI
  Groups: Patients diagnosed with suspected glioma scheduled for brain MRI; Patients with (suspected) glioma
Device: X-ray (optional) — Optional X-ray scan to assess the safety for undergoing an MR examination.
Combination Product: Additional contrast injection — Contrast agent administration for the additional 7T scan (optional).
  Groups: Patients diagnosed with suspected glioma scheduled for brain MRI; Patients with (suspected) glioma
Other: Question list — Questionnaire for contra-indications for an MR examination.

SUMMARY:
A glioma is a primary brain tumor in adults that is characterized by a highly variable, but overall poor survival. The optimal timing of treatment is in part determined by the expected biological behavior of the tumor. At present the expected biological behavior, determined by the tumor genotype, can only be determined by tissue analysis, which requires brain surgery. Non-invasive and improved diagnostic methods are sought to obtain insight into the molecular profile of the tumor and the expected biological behavior to avoid surgery performed solely for diagnostic purposes. Vascularization is an important aspect of the biological behavior of a primary brain tumor. Tumor vascularization characteristics can be assessed by Magnetic Resonance Imaging (MRI), but with the currently available technology this can only be achieved with unacceptably long scan times. In this proposal, the investigators will develop and optimize a novel MRI protocol to gather a large set of quantitative vascularization parameters within an acceptable scan time. The hypothesis is that from such a 'vascular signature' the tumor genotype can be inferred by means of machine learning.

DETAILED DESCRIPTION:
Objective of the study:

The primary objective is to develop and clinically validate a fast multi-parametric MRI acquisition technique, for non-invasive and comprehensive characterization of the tumor's vascularization, 'vascular signature mapping', at 3 Tesla (3T) and 7 Tesla (7T) MRI.

The secondary objective is to limit difficult and time-consuming visual interpretation of the acquired vascular information by developing a computer-aided diagnostic algorithm that automatically and accurately predicts the brain tumor genotype from the vascular signature maps.

Study design:

The study 'Vascular Signature Mapping for Brain Tumor Genotypes' is a multi-center observational diagnostic study, which consists of two parts. The first part of this study aims to develop and optimize a new MRI protocol that will exploit the effect of contrast agent on the MRI signal to infer information on the vascular properties of a tumor. It combines scans during the pre-contrast injection phase, the dynamic phase during and right after contrast agent injection, as well as the quasi static post-contrast phase. This research will focus on studying the optimal way of encoding the vascular architecture into the MRI signal and the decoding approach, In addition, the image processing methodology will be optimized. The second part of this study is a proof-of-concept clinical study. This part aims to link the vascular parameters with molecular profiles of tumors by using the collected data for the development of machine learning algorithms for predicting the tumor's genotype based on its vascular signature.

Study population:

The study population consists of 3 cohorts, all aged over 18 years, able to provide written informed consent and without contraindications for contrast-enhanced MRI. The first cohort, for development and optimization of the protocol, consists of 60 patients scheduled for brain MRI as part of their standard clinical diagnostic procedure and in whom contrast agent (CA) administration is part of their standard radiological assessment. These patients do not necessarily have a brain tumor as the purpose here is to develop and evaluate the vascular signature mapping sequence in general. The second cohort consists of 20 glioma patients in whom the vascular signature mapping sequence is tested and for a direct comparison between 3T and 7T MRI, where the 3T scan is an extension of the diagnostic care and the additional 7T scan is optional. The third cohort, for the clinical proof-of-concept study, consists of 100 adult patients referred for biopsy or surgery of suspected glioma.

Primary study parameters/outcome of the study:

The endpoint of the first part of the study is a novel MRI protocol for characterization of the vessel architecture, assessed with respect to the signal-to-noise ratio (SNR) and the ability to obtain vascular Information. The main parameters that will be used for characterization of the vasculature are physiological parameters including the vessel architecture, cerebral blood volume (CBV), cerebral blood flow (CBF), mean transit time (MTT), and oxygenation level.

The main study end point of the second part of the study is the accuracy of automatic classification of the tumor's genotype. The accuracy of the new method will be compared to the current state-of-the-art reference method based on conventional MRI.

Secondary study parameters/outcome of the study:

Baseline characteristics of subjects (including age, sex, Karnofsky performance status, tumor histology, molecular parameters (1p/19q, Isocitrate Dehydrogenase (IDH1/2) and 06-Methylguanine-DNA Methyltransferase (MGMT) status), tumor location, supportive and antitumor treatment). In addition, the outcome (e.g. mortality, tumor progression, radiation necrosis, functioning of patients) will be used as study parameter. The outcome will be determined from the follow-up scans after 3 and 6 months, where the criterion for progression or pseudo-progression is determined by the outcome of the scan.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

For the first cohort, the additional burden will not be substantial for the participant. The additional scan time will not exceed 10 minutes and therefore the impact on the patient will be limited. For the second and third cohort, the additional burden includes a prolonged MRI examination at a clinical MRI scanner (3T) and an optional additional examination at 7T MRI including additional CA injection. The ultrahigh field 7T MRI system is commonly used for research and no serious adverse events have been reported. Patients participating in this study will have no personal benefit; their participation aids in the development of a novel MRI method for the non-invasive determination of the tumor's molecular profile. Moreover, there is a small chance that the additional 7T MRI scan would provide more Information on the status of the disease in the participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for brain MRI with contrast injection as part of the clinical diagnostic procedure (cohort 1)
* Patients diagnosed with suspected glioma scheduled for brain MRI as part of the clinical diagnostic procedure (cohort 2)
* Patients with (suspected) glioma referred for tumor biopsy or resection (cohort 3)
* Age ≥ 18 years (all cohorts)
* Signed informed consent (all cohorts)

Exclusion Criteria:

* Subjects with contra-indications for an MRI exam
* Subjects with reduced kidney function because of the risk on developing nephrogenic systemic fibrosis (NSF) under gadolinium-based contrast injection
* Subjects with pregnancy
* Subjects undergoing a clinical protocol that requires scanning during CA injection (cohort 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first cohort, for protocol development and optimization, consists of 60 patients scheduled for brain MRI as part of their standard clinical diagnostic procedure and in whom contrast administration is part of their standard radiological assessment. These patients do not necessarily have a brain tumor as the purpose is to develop and evaluate the vascular signature mapping sequence in general. The second cohort consists of 20 glioma patients in whom the vascular signature mapping sequence is tested and for a direct comparison between 3T and 7T MRI, where the 3T scan is an extension of the diagnostic care and the additional 7T scan is optional. The third cohort, for the clinical proof-of-concept study, consists of 100 adult patients referred for biopsy or surgery of suspected glioma.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Optimized MR protocol | 6 months
  MR protocol optimized for SNR and the ability to obtain vascular information
Vessel architecture | 4 years
  Structure of vessels and tortuosity
Cerebral blood volume | 4 years
  To characterize the tumor's vasculature
Cerebral blood flow | 4 years
  To characterize the tumor's vasculature
Transit time parameters | 4 years
  Timing parameters used to characterize the tumor vasculature
Vascular oxygenation level | 4 years
  Oxygen-related parameters that describe the tumor's vasculature

SECONDARY OUTCOMES:
Basic subject characteristics | 4 years
  Age, gender, KPS performance score
Tumor histology | 4 years
  Structural information about the tumor, cell type and architectural pattern
Tumor molecular parameters | 4 years
  IDH mutation, MGMT status
Treatment information | 4 years
  Radiotherapy dose, chemotherapy scheme
Tumor progression scored on follow-up MR scan | 4 years
  Assessment of tumor progression versus pseudo-progression based on scoring of follow-up MR scans by an experienced physician.
Radiation necrosis evaluated on follow-up MR scan | 4 years
  Assessment based on evaluation of follow-up MR scans by an experienced physician.
Mortality | 4 years
  Survival time and occurrence of death
KPS score at follow-up of 3 and 6 months | 4 years
  Performance score providing information about the functioning of patients

CONTACTS AND LOCATIONS:
Overall Officials: Matthias JP van Osch, Prof Dr Ir, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smits M, van den Bent MJ. Imaging Correlates of Adult Glioma Genotypes. Radiology. 2017 Aug;284(2):316-331. doi: 10.1148/radiol.2017151930. PMID 28723281
- [Background] van den Bent MJ, Smits M, Kros JM, Chang SM. Diffuse Infiltrating Oligodendroglioma and Astrocytoma. J Clin Oncol. 2017 Jul 20;35(21):2394-2401. doi: 10.1200/JCO.2017.72.6737. Epub 2017 Jun 22. PMID 28640702
- [Background] Killela PJ, Pirozzi CJ, Healy P, Reitman ZJ, Lipp E, Rasheed BA, Yang R, Diplas BH, Wang Z, Greer PK, Zhu H, Wang CY, Carpenter AB, Friedman H, Friedman AH, Keir ST, He J, He Y, McLendon RE, Herndon JE 2nd, Yan H, Bigner DD. Mutations in IDH1, IDH2, and in the TERT promoter define clinically distinct subgroups of adult malignant gliomas. Oncotarget. 2014 Mar 30;5(6):1515-25. doi: 10.18632/oncotarget.1765. PMID 24722048
- [Background] Louis DN, Perry A, Reifenberger G, von Deimling A, Figarella-Branger D, Cavenee WK, Ohgaki H, Wiestler OD, Kleihues P, Ellison DW. The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary. Acta Neuropathol. 2016 Jun;131(6):803-20. doi: 10.1007/s00401-016-1545-1. Epub 2016 May 9. PMID 27157931
- [Background] Holash J, Maisonpierre PC, Compton D, Boland P, Alexander CR, Zagzag D, Yancopoulos GD, Wiegand SJ. Vessel cooption, regression, and growth in tumors mediated by angiopoietins and VEGF. Science. 1999 Jun 18;284(5422):1994-8. doi: 10.1126/science.284.5422.1994. PMID 10373119
- [Background] Fischer I, Gagner JP, Law M, Newcomb EW, Zagzag D. Angiogenesis in gliomas: biology and molecular pathophysiology. Brain Pathol. 2005 Oct;15(4):297-310. doi: 10.1111/j.1750-3639.2005.tb00115.x. PMID 16389942
- [Background] Koeller KK, Rushing EJ. From the archives of the AFIP: Oligodendroglioma and its variants: radiologic-pathologic correlation. Radiographics. 2005 Nov-Dec;25(6):1669-88. doi: 10.1148/rg.256055137. PMID 16284142
- [Background] Law M, Young RJ, Babb JS, Peccerelli N, Chheang S, Gruber ML, Miller DC, Golfinos JG, Zagzag D, Johnson G. Gliomas: predicting time to progression or survival with cerebral blood volume measurements at dynamic susceptibility-weighted contrast-enhanced perfusion MR imaging. Radiology. 2008 May;247(2):490-8. doi: 10.1148/radiol.2472070898. Epub 2008 Mar 18. PMID 18349315
- [Background] Caseiras GB, Chheang S, Babb J, Rees JH, Pecerrelli N, Tozer DJ, Benton C, Zagzag D, Johnson G, Waldman AD, Jager HR, Law M. Relative cerebral blood volume measurements of low-grade gliomas predict patient outcome in a multi-institution setting. Eur J Radiol. 2010 Feb;73(2):215-20. doi: 10.1016/j.ejrad.2008.11.005. Epub 2009 Feb 6. PMID 19201123
- [Background] Grobner T. Gadolinium--a specific trigger for the development of nephrogenic fibrosing dermopathy and nephrogenic systemic fibrosis? Nephrol Dial Transplant. 2006 Apr;21(4):1104-8. doi: 10.1093/ndt/gfk062. Epub 2006 Jan 23. No abstract available. PMID 16431890
- [Background] van der Voort SR, Incekara F, Wijnenga MMJ, Kapas G, Gardeniers M, Schouten JW, Starmans MPA, Nandoe Tewarie R, Lycklama GJ, French PJ, Dubbink HJ, van den Bent MJ, Vincent AJPE, Niessen WJ, Klein S, Smits M. Predicting the 1p/19q Codeletion Status of Presumed Low-Grade Glioma with an Externally Validated Machine Learning Algorithm. Clin Cancer Res. 2019 Dec 15;25(24):7455-7462. doi: 10.1158/1078-0432.CCR-19-1127. Epub 2019 Sep 23. PMID 31548344